CLINICAL TRIAL: NCT04386161
Title: Static and Dynamic Balance Changes After a Scheduled Exercise Program in Children With Dyslexia
Brief Title: Static and Dynamic Balance in Children With Dyslexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Kardelen Gencer Atalay, Principal Investigator, Marmara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09.2017.672
Record Dates: First submitted 2020-05-05; First posted 2020-05-13 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Dyslexia
Keywords: Dyslexia; Balance; Exercise Program
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Intervention Model Description: Children, aged between 8 and 11 years, with clinical dyslexia diagnosed by a child and adolescent psychiatrist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with dyslexia (Experimental): Children, aged between 8 and 11 years, with clinical dyslexia diagnosed by a child and adolescent psychiatrist
  Interventions: Other: Scheduled exercise program

INTERVENTIONS:
Other: Scheduled exercise program — 45 minutes of stretching, strengthening, and balance-coordination exercises and 20 minutes of balance training on the Balance Master® device twice a week for six weeks

SUMMARY:
Dyslexia is described as a learning disability with a neurological origin. It is a widespread disease, characterized by difficulties in recognition of words, spelling, and decoding.

Postural balance is the ability to control the center of gravity (CoG) on the support base. This control starts to appear at the beginning of the 15th months of life and reaches its maximum capacity at around 12 years with the maturation of visual, vestibular, and somatosensory systems. Static balance defines the postural control state in the maintaining position, while dynamic balance represents it during movement. Static and dynamic balance has been widely investigated and found to be impaired in different pediatric disorders such as cystic fibrosis, cerebral palsy, and spina bifida. There is also apparent evidence of deteriorated balance in children with dyslexia. Although quite a number of studies investigated balance impairment in individuals with dyslexia, only one study was interested in the effects of a postural training program and found significant improvements. That study addressed such improvements to brain plasticity, however, did not investigate the reading performance simultaneously. The aim of this study was to demonstrate the changes in static and dynamic balance, reading performance, and quality of life after a six week after a scheduled exercise program in children with dyslexia.

DETAILED DESCRIPTION:
Dyslexia is described as a learning disability with a neurological origin. It is a widespread disease, characterized by difficulties in recognition of words, spelling, and decoding. It is an unexpected and permanent failure in gaining reading skills in the individual who have sufficient intelligence, socio-cultural opportunities, and education, according to the World Health Organization. The diagnosis can be made by a child and adolescent psychiatrist clinically or with the Diagnostics and Statistical Manual of mental disorders (DSM-5). The prevalence of dyslexia varies between 2-10%, and it is seen 3-4 times more in men than in women.

Postural balance is the ability to control the center of gravity (CoG) on the support base. This control starts to appear at the beginning of the 15th months of life and reaches its maximum capacity at around 12 years with the maturation of visual, vestibular, and somatosensory systems. Static balance defines the postural control state in the maintaining position, while dynamic balance represents it during movement. Static and dynamic balance has been widely investigated and found to be impaired in different pediatric disorders such as cystic fibrosis, cerebral palsy, and spina bifida. There is also apparent evidence of deteriorated balance in children with dyslexia. Frankle and Levinson suggested that there is a cerebellar-vestibular disorder in people with dyslexia for the first time in 1973. They found that 97% of 115 children with dyslexia abnormal neurological findings such as positive Romberg test, walking difficulty, speech disorder, or hypotonia. After then, Rae et al. reported that the right frontal lobe of the cerebellum was smaller, and there were distinct biochemical changes on the temporoparietal lobe in dyslexic individuals compared to healthy controls. Moe-Nilssen et al. showed that dyslexic children have impairment in both balance and gait ability. Barela et al. claimed that writing and learning disorders in dyslexia were associated with cerebellum. Patel et al. found that postural instability was related to the severity of dyslexia. Quercia et al. gave postural exercise treatment to the dyslexics, then examined their postural stability after a vibrational stimulation. The length and speed of CoG were shown to be significantly higher in untreated dyslexic patients compared to the treated dyslexics and the non-dyslexic group.

Although quite a number of studies investigated balance impairment in individuals with dyslexia, only one study was interested in the effects of a postural training program and found significant improvements. That study addressed such improvements to brain plasticity, however, did not investigate the reading performance simultaneously. The aim of this study was to demonstrate the changes in static and dynamic balance, reading performance, and quality of life after a six week after a scheduled exercise program in children with dyslexia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with dyslexia by a child and adolescent psychiatrist
* WISC R test result in IQ> 85

Exclusion Criteria:

* Having hyperactivity disorder according to DSM-5
* Having a neuromuscular disease, skeletal anomaly, or vision and hearing problem
* Using an antipsychotic drug

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Static Balance Assessment | Day 0
  Postural sway velocities on the firm and foam surfaces with eyes opened and closed conditions of Modified Clinical Test of Sensory Interaction on Balance (mCTSIB) test
Static Balance Assessment | Week 6
  Postural sway velocities on the firm and foam surfaces with eyes opened and closed conditions of Modified Clinical Test of Sensory Interaction on Balance (mCTSIB) test

SECONDARY OUTCOMES:
Dynamic Balance Assessment, Reaction time | Day 0
  Reaction time of Limits of Stability (LOS) test
Dynamic Balance Assessment, Reaction time | Week 6
  Reaction time of Limits of Stability (LOS) test
Dynamic Balance Assessment, Movement time | Day 0
  Movement time of Limits of Stability (LOS) test
Dynamic Balance Assessment, Movement time | Week 6
  Movement time of Limits of Stability (LOS) test
Dynamic Balance Assessment, Endpoint excursion | Day 0
  Endpoint excursion of Limits of Stability (LOS) test
Dynamic Balance Assessment, Endpoint excursion | Week 6
  Endpoint excursion of Limits of Stability (LOS) test
Dynamic Balance Assessment, Maximum excursion | Day 0
  Maximum excursion of Limits of Stability (LOS) test
Dynamic Balance Assessment, Maximum excursion | Week 6
  Maximum excursion of Limits of Stability (LOS) test
Dynamic Balance Assessment, Direction control | Day 0
  Direction control of Limits of Stability (LOS) test
Dynamic Balance Assessment, Direction control | Week 6
  Direction control of Limits of Stability (LOS) test
Reading Performance | Day 0
  The number of correct and total words
Reading Performance | Week 6
  The number of correct and total words
Pediatric Quality of Life Inventory Scale | Day 0
  There are 23 questions in this scale and 5 options for each question, it takes a short time to complete and contains questions about physical, social, emotional and school functionality. For the questions, zero means that the person never had a problem, and four means that the person always has a problem.
Pediatric Quality of Life Inventory Scale | Week 6
  There are 23 questions in this scale and 5 options for each question, it takes a short time to complete and contains questions about physical, social, emotional and school functionality. For the questions, zero means that the person never had a problem, and four means that the person always has a problem.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Karadag Saygi, Study Director — Marmara University
Locations (1):
- Kardelen Gencer Atalay, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No